CLINICAL TRIAL: NCT03618888
Title: Pedagogical Aspects on Education in Basic Life Support: A Cluster Randomized Trial on Effectiveness, Comparing Different Educational Methods for Adults in the Society of Sweden.
Brief Title: Pedagogical Aspects on Training in Basic Life Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Boras (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Principal Investigator, Helene Bylow, RNAN, Master of Pedagogy, PhD Student, University of Gothenburg, University of Boras, University of Boras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Johan Herlitz
Record Dates: First submitted 2018-07-21; First posted 2018-08-07 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Basic Life Support
Keywords: Out-of-Hospital Cardiac arrest; Cardiopulmonary Resuscitation; Automated External Defibrillator; Self-learning; Basic Life Support
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Parallel Assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instructor-led training (Active Comparator): Instructor-led training contents a supervised practical training for BLS, facilitated by a certified instructor.
  Interventions: Other: Instructor-led training
- Self-learning training (Experimental): Self-learning training is self-directed and contents practical training for BLS
  Interventions: Other: Self-learning training

INTERVENTIONS:
Other: Instructor-led training — The Instructor-led training contents a supervised practical training with a standard kit for training in BLS
  Arms: Instructor-led training
Other: Self-learning training — The self-learning training contents a standard kit for self-directed training in BLS
  Arms: Self-learning training

SUMMARY:
Cardio vascular disease (CVD) including out-of-hospital cardiac arrest (OHCA) is still the leading cause of death in a global perspective. Start of cardiopulmonary resuscitation (CPR) with automated external defibrillator (AED) may double or quadruple survival. Scientific research on education in Basic Life Support (BLS) in the society is active in different part of Europe but low in Sweden. The aim of this study is to investigate the effectiveness and retention after different training interventions in BLS and willingness to act in a real-life cardiac arrest situation in the society of Sweden, based on European Resuscitation Council (ERC) guidelines. This is an experimental cluster randomized trial, including participants from a BLS education project in Sweden.

DETAILED DESCRIPTION:
Introduction: The single most important factor for survival from sudden cardiac arrest (SCA) is to minimize the time from cardiac arrest to cardiopulmonary resuscitation (CPR) and to provide an electric chock through the heart with an automated external defibrillator (AED). Early start with CPR-AED increases the chance of survival two to four times. It is therefore important that as many people as possible have knowledge to quickly identify SCA and to start CPR-AED.

In this research, education efforts are directed for the adult public at workplaces in Sweden. The Investigator have designed an intervention in accordance to guidelines from European Resuscitation Council (ERC) and the Swedish national education for Basic Life Support (BLS).

This is a cluster randomized trial primarily comparing in the first study, instructor-led training as the control group and self-learning training as the experimental group. In the second study the Investigator plan to compare a preparatory web-education on CVD before the BLS training versus no web-education before the BLS. The Investigator have conducted quality tests on practical skills on BLS, administered questionnaires to the participants about theoretical knowledge, self-assessed confidence and willingness to act in a real-life SCA situation. It is crucial to be able to identify factors that affect knowledge and retention after BLS training and the willingness to intervene in an acute situation.

Background: With modern IT technology, several different options and learning strategies are available. At the same time pedagogical thoughts have emerged on learning. Education can be instructor-led or self-directed and with preparatory courses for theoretical knowledge. The quality of BLS skills and theoretical knowledge can be measured through validated instruments. Against this background, the research goal is to identify how the study can improve retention and which training methods for BLS that should be recommended for the public in the future.

Objectives: The overall objective is to increase survival from OHCA. The aim is to identify factors that affect retention and contributes to intended practical skills, theoretical knowledge and willingness to act after BLS training and whether these goals are affected by the type of training intervention.

Hypothesis: The main hypothesis is that retention of practical skills after BLS training is affected by the type of educational intervention. The hypothesis in the first study is that an instructor present at the time of training have a positive impact on retention six months after the intervention compared to self-directed training. In the second study the hypothesis is that a preparatory web-education on CVD before the BLS has a positive impact on retention six months after intervention compared to no web-education.

Questions: The Primary question is which intervention is most effective for the total score and contributes to intended practical skills and adherence to protocol, the BLS algorithm, six months after the intervention. Secondary questions deal with if other variables such as practical skills, theoretical knowledge, self-assessed confidence and willingness to intervene in a SCA situation are affected when comparing each intervention both direct after and six months after training.

Method: Voluntary, participants from a BLS project at workplaces in Sweden have been included. The participants have been randomized from a randomization list and organized for the study, from an independent coordinator. After training and at six months, a quantitative approach and data collection measured the quality of practical skills in a simulated SCA scenario, on a Laerdal Resusci Anne manikin, connected to the PCSkillReporting system. The assessor was blinded for the type of training intervention. At data collection, the variables were structured according to a modified international quality test, Cardiff Test of basic life support and automated external defibrillation (Cardiff Test) that scored adherence to the treatment algorithm and practical skills. The modified Cardiff Test included 19 variables with a total score of 70 points. A questionnaire scored theoretical knowledge, self-assessed confidence and willingness to act in a real-life situation. At the practical quality tests, the total score was the primary endpoint with other individual variables as the secondary endpoint.

Study population: Strategic sampling was used to include participants from different workplaces in a number of counties in Sweden.

Planned Studies: 1) Self-learning training versus Instructor-led training. 2) A preparatory web-education on CVD before the BLS training versus no web-education before the BLS training. 3) A register study on bystander activity 4) Instructor-led training versus subgroups of training from the BLS intervention project.

Statistics: All statistical analyses will be analysed in SASforwindows and calculated on a cluster level with an alpha level of five percent.

Ethical considerations: Ethical principles for research are carefully considered in the research process. Ethical vetting from Ethical Review of Research, involving Humans is approved (Regional Ethical Review Board in Gothenburg, diaries number 134-14) and Guidelines from the Swedish Research Council, Good Research Practice is actively used. Information has been given both individually to all participants and to the working places. All participant had to read and sign a personal consent form before participating. The result will be published according to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion criteria

* Adults in society over eighteen years old
* Working at workplaces outside hospital
* Without training in BLS or within the past five years
* A completed and signed consent form.

Exclusion criteria

* Participants younger than 18 years old
* Undergone training on BLS within the past five years
* Working at hospital as health care personnel
* Do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2623 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Total score from Cardiff Test for retention at 6 months | 6 months after intervention
  Total score from the modified instrument Cardiff Test on the participants individual practical skills and adherence to the Basic Life Support algorithm in retention-test at six months after intervention.

SECONDARY OUTCOMES:
Individual quality variables from PC SkillReporting System at baseline and at retention at 6 months. | 0 days + 6 months later
  Individual quality variables from the instrument and data program PC SkillReporting system on the participants quality on practical skills for Basic Life Support at baseline as post-test direct after intervention, as retention-test at six months later and as a change in quality of Basic Life Support
Self-assessed theoretical knowledge from questionnaires at baseline and retention at 6 months | 0 days + 6 months later
  Self-assessed theoretical knowledge with data collected from the participants individual questionnaires at baseline as post-test direct after intervention and as retention-test at six months later.
Self-assessed confidence from questionnaires at baseline and retention at 6 months | 0 days + 6 months later
  Self-assessed confidence after the intervention with data collected from the participants individual questionnaires at baseline and retention at six months later.
Self-assessed willingness from questionnaires at baseline and retention at 6 months | 0 days + 6 months later
  Self-assessed willingness to act in a real-life sudden cardiac arrest situation with data collected from the participants individual questionnaires at baseline and retention at six months later.
Theoretical knowledge on cardio vascular disease, symptoms and first actions from questionnaires at baseline and retention at 6 months | 0 days + 6 months later
  Theoretical knowledge on cardio vascular disease, first actions and healthy life style factors with data collected from the participants individual questionnaires at baseline and retention at six months later. Secondary Outcome for study 2) A preparatory web-education on CVD before the BLS training versus no web-education before the BLS training.
Self-assessed experience on learning outcome at baseline and retention at 6 months | 0 days + 6 months later
  Self-assessed experience on the participants individual learning outcome at baseline and retention at six months with data collected from the participants individual questionnaires at baseline and retention at six months later. Secondary Outcome for study 4) Instructor-led training versus subgroups of training from the BLS intervention project.

CONTACTS AND LOCATIONS:
Overall Officials: Johan D Herlitz, Professor, Principal Investigator — University of Borås Sweden
Locations (1):
- University of Borås Sweden, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will be analysed and published on group level only

REFERENCES:
- [Derived] Bylow H, Karlsson T, Lepp M, Claesson A, Lindqvist J, Svensson L, Herlitz J. Learning Outcome After Different Combinations of Seven Learning Activities in Basic Life Support on Laypersons in Workplaces: a Cluster Randomised, Controlled Trial. Med Sci Educ. 2020 Nov 18;31(1):161-173. doi: 10.1007/s40670-020-01160-3. eCollection 2021 Feb. PMID 34457876
- [Derived] Bylow H, Karlsson T, Claesson A, Lepp M, Lindqvist J, Herlitz J. Self-learning training versus instructor-led training for basic life support: A cluster randomised trial. Resuscitation. 2019 Jun;139:122-132. doi: 10.1016/j.resuscitation.2019.03.026. Epub 2019 Mar 26. PMID 30926451